CLINICAL TRIAL: NCT01376011
Title: Hypoxia-inducible Transcription Factor 1 (HIF-1) in Vascular Aging
Brief Title: Modulation of Cerebral Blood Flow Using Quercetin, a Nutritional Supplement
Acronym: Quercetin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Farzaneh Sorond, Principle Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1 K23AG030967-01A1-2; 1K23AG030967-01A1 (NIH)
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Stroke; Problem of Aging
Keywords: quercetin; brain blood flow; aging; memory
MeSH Terms: conditions — Stroke | interventions — Quercetin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- healthy young (Experimental)
  Interventions: Dietary Supplement: quercetin/placebo
- healthy old (Experimental)
  Interventions: Dietary Supplement: quercetin/placebo

INTERVENTIONS:
Dietary Supplement: quercetin/placebo — Quercetin 500mg once per day versus placebo

SUMMARY:
The purpose of this study is to find out if quercetin can increase blood levels of hypoxia-inducible transcription factor 1 (HIF-1 protein) and to see if there is a corresponding increase in blood flow to the brain.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers between the ages of 18-75 years old

Exclusion Criteria:

* subjects taking vasoactive medications
* hypertension or vascular disease
* asthma
* smokers
* pregnant women
* cancer
* diabetes mellitus
* history of seizures
* history of stroke or head trauma
* subjects taking digoxin, cyclosporine,felodipine, estradiol, or quinolone antibiotics
* poor transcranial Doppler insonation windows

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Define change from baseline levels of HIF-1 concentration and 3 of its regulated proteins after 6 months of quercetin (versus placebo) dietary intake. | 6 months
  Baseline and 6 month blood samples will be analyzed for levels of HIF-1, VEGF, EPO, and NOS
Determine change from baseline brain blood flow after 6 months of quercetin (versus placebo) dietary intake. | 6 months
  Determine cerebral vasomotor reactivity response to 6 months of quercetin intake by measuring changes in middle cerebral artery (MCA) blood flow velocity in response to changes in end-tidal CO2, and assess neurovascular coupling by measuring changes in MCA flow velocity in response to neuropsychological tasks.

SECONDARY OUTCOMES:
Define change from baseline performance in a battery of cognitive tasks after 6 months of quercetin (versus placebo) dietary intake. | 6 months
  Assess effects of 6 months of quercetin intake on cognitive function using a cognitive battery designed to asses both memory and executive function.

CONTACTS AND LOCATIONS:
Overall Officials: Farzaneh Sorond, mD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States